CLINICAL TRIAL: NCT07133867
Title: Evaluation of Artificial Intelligence in Planning the Treatment for Cases With Missing Upper Lateral Incisors (A Diagnostic Accuracy Pilot Study)
Brief Title: AI-Guided Treatment Planning in Orthodontic Patients With Missing Upper Lateral Incisors
Acronym: SMILE-AI
Status: Active, not recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Malak Mohsen Ahmed Elagramy, Master's Candidate in Orthodontics" Faculty of Oral and Dental Medicine, Cairo University, Cairo University
Other Study IDs: ORTH 7-1-3
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Orthodontic Treatment Planning; Congenitally Missing Maxillary Lateral Incisors
Keywords: Artificial Intelligence; orthodontics; missing lateral incisor; treatment planning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This pilot study aims to evaluate the diagnostic accuracy of artificial intelligence (AI) in orthodontic treatment planning for patients with congenitally missing upper lateral incisors. The study compares AI-generated treatment recommendations with decisions made by experienced orthodontists regarding two main treatment options: space closure and prosthetic replacement. Orthodontic records, including intraoral and extraoral photographs, panoramic radiographs, and cephalometric analyses, will be collected for each case. Two orthodontists with over 10 years of clinical experience will independently evaluate each case using a treatment decision checklist with predefined cutoff points. AI predictions will then be compared to orthodontists' consensus decisions to determine agreement rates and accuracy. The findings will provide insight into the potential role of AI in supporting complex orthodontic decision-making.

DETAILED DESCRIPTION:
Management of congenitally missing maxillary lateral incisors is a frequent clinical challenge in orthodontics, often sparking debate among practitioners regarding the optimal treatment approach. The two primary treatment modalities are orthodontic space closure, in which adjacent teeth (usually canines) are moved into the lateral incisor position, and space opening followed by prosthetic replacement, typically with dental implants or bridges. Each option has distinct advantages and limitations in terms of esthetics, occlusion, periodontal health, and long-term stability, and the decision is influenced by multiple clinical, biological, esthetic, and patient-specific factors.

Artificial intelligence (AI), particularly through machine learning algorithms, has demonstrated high accuracy in other controversial orthodontic decision-making scenarios, such as extraction vs. non-extraction treatment and surgical vs. camouflage approaches. However, its application to lateral incisor agenesis treatment planning has not been thoroughly investigated.

This pilot diagnostic accuracy study will evaluate the performance of an AI-based decision support system in recommending treatment plans for cases with missing maxillary lateral incisors. A dataset of anticipated 100 cases will be compiled, consisting of pre-treatment records including intraoral and extraoral photographs, panoramic radiographs, and cephalometric analyses. two experienced orthodontists will independently review unfinished cases and make a treatment decision-space closure, space opening with prosthetic replacement, or undecided-using a standardized cutoff-points checklist. For finished cases, both pre- and post-treatment records will be analyzed.

A consensus decision will be established when at least two orthodontists agree; if disagreement persists, a third orthodontist will finalize the decision. AI predictions will be compared with orthodontists' consensus decisions to assess diagnostic accuracy, sensitivity, specificity, and agreement rates. This study aims to explore the feasibility of integrating AI tools into complex orthodontic decision-making and to establish a foundation for larger-scale clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with unilateral or bilateral congenitally missing maxillary lateral incisors (confirmed by panoramic radiograph).
* Availability of complete diagnostic records: intraoral photographs, extraoral photographs, cephalometric radiograph, and panoramic radiograph.
* Cases either finished (completed orthodontic treatment) or unfinished (under treatment).
* No prior prosthetic replacement for the missing lateral incisors before initial orthodontic planning.

Exclusion Criteria:

* Patients with craniofacial syndromes or cleft lip/palate.
* Cases with incomplete or poor-quality diagnostic records.
* History of previous orthodontic treatment unrelated to the current missing lateral incisor case.
* Multiple missing teeth outside the upper lateral incisor region that could affect treatment planning.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Orthodontic patients with confirmed diagnosis of congenital absence of one or both maxillary lateral incisors, treated or being treated at the Faculty of Oral and Dental Medicine, Cairo University, and collaborating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of AI in Orthodontic Treatment Planning for Missing Maxillary Lateral Incisors | Within 6 months from case assessment
  The percentage agreement between AI-generated treatment decisions (space closure vs. space opening) and the consensus decisions of experienced orthodontists, based on standardized case records including intraoral photographs, cephalometric radiographs, and panoramic radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Professor (Associate), Study Director — orthodontic department-cairo university
Locations (1):
- Faculty of Oral and Dental Medecine -Cairo University, Cairo, Manial, Egypt